CLINICAL TRIAL: NCT06759688
Title: Role of Low Carbohydrate Nutrient in Healing of Infected Diabetic Foot
Acronym: LCN
Status: Completed | Type: Observational
Sponsor: Sarah Magdy Abdelmohsen (Other)
Responsible Party: Sponsor-Investigator, Sarah Magdy Abdelmohsen, Principle investigator, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Other Study IDs: AswanUH7
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Carbohydrate Ingestion
Keywords: Diabetic foot wound infections,; Diabetic foot ulcer,; low carbohydrate dietary approaches.
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic foot infection with carbohydrates restriction group: It involving patients with diabetic foot infections. The patients were divided into two groups of patients. The first group committed to not eating carbohydrates in food. The second group ate their daily routine and did not adhere to the carbohydrate's restriction. The diabetic food infection classified from mild, moderate and sever, as per the Infectious Diseases Society of America (IDSA) Infection Severity Classification.
  Interventions: Behavioral: Carbohydrates restriction
- diabetic foot infection without carbohydrates restriction: It involving patients with diabetic foot infections. The patients were divided into two groups of patients. The first group committed to not eating carbohydrates in food. The second group ate their daily routine and did not adhere to the carbohydrate's restriction. The diabetic food infection classified from mild, moderate and sever, as per the Infectious Diseases Society of America (IDSA) Infection Severity Classification.

INTERVENTIONS:
Behavioral: Carbohydrates restriction — Patients followed a low carbohydrate dietary approach (LCDs). It means lower than 130 grams carbohydrates per day with special restriction restrictions on:
  * Artificial sugars (e.g., sweets, baked goods, pasta, bread).
  * Also, rice, butter made from vegetable oils and all types of oils except olive oil.
  They were allowed:
  * All types of fresh fruits and vegetable.
  * Boiled potatoes.
  Other Names: diabetic foot infection with low carbohydrates diet
  Groups: diabetic foot infection with carbohydrates restriction group

SUMMARY:
A low-carbohydrate diet, when combined with standard wound care and diabetes management, appears to accelerate the healing of infected diabetic foot, improve blood glucose control, reduce systemic inflammation and promoting overall patient recovery. This approach could be considered a beneficial adjunct therapy in the treatment of diabetic foot infections.

DETAILED DESCRIPTION:
The research was a case control study. It conducted prospectively from January 2019 to December 2023 in the surgery department of Aswan university hospital. It involving patients with diabetic foot infections. The patients were divided into two groups of patients. The first group committed to not eating carbohydrates in food. The second group ate their daily routine and did not adhere to the carbohydrate's restriction. The diabetic food infection classified from mild, moderate and sever, as per the Infectious Diseases Society of America (IDSA) Infection Severity Classification.

ELIGIBILITY:
Inclusion Criteria:

Patients complained of diabetic foot infections graded 0 to 4 with absent signs of ischemia.

Exclusion Criteria:

Patients with foot gangrene grade 5 The presence of foot ischemia Those who refused to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients complained of diabetic foot infections graded 0 to 4 with absent signs of ischemia.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the wound size and healing | 3-6 months
  Wound healing rate (%) = [ (Initial wound size - Wound size after 1 week) / (Initial wound size)] × 100

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol